CLINICAL TRIAL: NCT05988528
Title: Clinical Study to Evaluate the Possible Efficacy of Nifuroxazide in Patient With Ulcerative Colitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mostafa Bahaa (Other)
Responsible Party: Sponsor-Investigator, Mostafa Bahaa, Teaching assisstant, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8/2023
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Mesalamine; nifuroxazide

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: double blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): Control group (Mesalamine group, n =30 ) who will receive 1 g mesalamine three times daily for 6 months
  Interventions: Drug: Mesalamine
- Nifuroxazide group (Active Comparator): Patients will receive 1 g mesalamine three times daily plus Nifuroxazide 200 mg two times daily for 6 months
  Interventions: Drug: Mesalamine; Drug: Nifuroxazide

INTERVENTIONS:
Drug: Mesalamine — Mesalamine, also known as 5-aminosalicylic acid (5-ASA), is a medication used to treat ulcerative colitis. It is usually used to induce or maintain remission of mildly to moderately active ulcerative colitis.
Drug: Nifuroxazide — Nifuroxazide is an oral antibiotic that has been approved as an effective antidiarrheal agent with no side effects in several gastrointestinal infections
  Arms: Nifuroxazide group

SUMMARY:
Ulcerative colitis (UC) is one of the most common types of chronic and non-specific inflammatory bowel diseases (IBD). It is characterized by cytokine-induced continuous and diffuse inflammatory infiltrations into the rectum's mucosa and extends proximally to the colon. Patients with UC predominantly have bloody diarrhea, abdominal pain, fecal urgency, and tenesmus, which extremely alters their quality of life.

Although the precise pathological mechanism of UC remains unclear, several studies have been outlined many factors that could involve in the pathogenesis of UC, including, but not limited to, initiation of the inflammatory response, disruption of oxidant/antioxidant status, dysregulation of the immune response, alteration of gut microbiota, and delaying epithelial barrier healing. Loss of intestinal barrier function and dysregulated immune response are the key events during colitis development

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Both male and female will be
* Mild and moderate UC patients diagnosed and confirmed by endoscope

Exclusion Criteria:

* Breast feeding
* Significant liver and kidney function abnormalities
* Colorectal cancer patients
* Other inflammatory bowel diseases (CD).
* Patients with severe UC
* Patients taking rectal or systemic steroids
* Patients taking immunosuppressives or biological therapies
* Addiction to alcohol and / or drugs
* Known allergy to the Fenofibrate

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-08-20 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the improvement in health-related quality of life | 6 months
  The IBDQ includes 32 questions, The questions are grouped into four categories: bowel symptoms (B), systemic symptoms (S), emotional function (E), and social function (SF). Response options are consistently presented as seven-point scales, scores range from 32-224

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, Egypt

REFERENCES:
- [Derived] AlRasheed HA, Abdallah MS, El-Khateeb E, Kamal M, Alrubia S, Alsegiani AS, Ahmed TI, Bahaa MM. A Randomized Controlled Pilot Study Evaluating the Safety and Efficacy of Nifuroxazide in Patients with Ulcerative Colitis. Drug Des Devel Ther. 2025 Jun 30;19:5539-5552. doi: 10.2147/DDDT.S522755. eCollection 2025. PMID 40620467